CLINICAL TRIAL: NCT03872752
Title: Development and Implementation of Food Literacy Workshops in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FL-HMO-CTIL
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lifestyle Risk Reduction; Health Behavior; Food Habits
MeSH Terms: conditions — Risk Reduction Behavior; Health Behavior; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This study includes a pre/post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lay leader training in FL intervention (Experimental): Community lay leaders from pre-existing community frameworks will undergo training in a manualized program that enables lay leaders to effectively disseminate food literacy skills through engaging visual and game-based tools in a food literacy workshop. Post training, lay leaders will implement the food literacy workshop in their communities.
  Interventions: Behavioral: FL lay leader training and workshop implementation

INTERVENTIONS:
Behavioral: FL lay leader training and workshop implementation — Intervention components will include a training course for community lay leaders, enabling them to acquire the skills to lead food literacy workshops. This includes raising their knowledge about nutrition recommendations and food labels, raisin self efficacy, and improving nutrition related organization and preparation skills.

SUMMARY:
Nutritional factors are responsible for 10% of the global health burden. In Israel, 31% of Jewish women and 52% of Arab women are obese. It is predicted that this generation will see increased cardiovascular disease (CVD) and decreased life expectancy. Sustained lifestyle changes including small changes in nutrition behavior, can substantially reduce the risk of CVD.

Eating habits are affected by different abilities, circumstances, and skill sets, however, most nutrition programs focus on nutrition facts, and less on skills that can help translate knowledge to positive health behaviors and health outcomes. In the last decade a new field has emerged, Food literacy (FL), which acknowledges the importance of addressing skills such as nutrition knowledge, competencies, self-efficacy, literacy and health literacy, so as to enable positive change in nutrition behaviors. Food literacy, in summary, is the capability to make healthy food choices in different contexts, settings and situations.

The proposed program seeks to improve nutrition behaviors in disadvantaged communities via a train-the-trainers program, that will provide community leaders with the tools necessary to disseminate FL skills through the framework of existing community social-structures.

DETAILED DESCRIPTION:
Nutritional factors are responsible for 10% of the global health burden. In Israel, 31% of Jewish women and 52% of Arab women are obese. Diabetes rates are rising in accordance with the rise in obesity. Because of these factors, it is predicted that this generation will see increased cardiovascular disease (CVD) and decreased life expectancy. Sustained lifestyle changes including small changes in nutrition behavior, can substantially reduce the risk of CVD.

Eating habits are affected by different abilities, circumstances, and skill sets, however, most nutrition programs focus on nutrition facts, and less on skills that can help translate knowledge to positive health behaviors and health outcomes. In the last decade a new field has emerged, Food literacy (FL), which acknowledges the importance of addressing skills such as nutrition knowledge, competencies, self-efficacy, literacy and health literacy, so as to enable positive change in nutrition behaviors. FL, in summary, is the capability to make healthy food choices in different contexts, settings and situations.

The proposed program seeks to improve nutrition behaviors in disadvantaged communities via a train-the-trainers program, that will provide community leaders with the tools necessary to disseminate food literacy skills through the framework of existing community social-structures.

In stage I of the study, community lay leaders from pre-existing community frameworks of Hebrew speaking communities and Arab lay leaders from East Jerusalem will undergo training in a manualized program that enables lay leaders to effectively disseminate FL skills through engaging visual and game-based tools. In stage II the lay leaders will implement the program in their communities.

ELIGIBILITY:
Inclusion Criteria:

* Women who are recognized leaders in the community will be included in training courses
* Participants for the Arab training program must speak and read Arabic
* Participants for the Hebrew-speaking training program must speak and read Hebrew

Exclusion Criteria:

- women who do not meet leadership criteria will be considered for training

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of lay-led workshops assessed by attendance rates | Throughout workshops, taking place throughout one year
  Attendance is monitored to calculate proportion of attendance of participants.
Feasibility of lay-led workshops assessed by number of implemented workshops by lay-leaders | six months after last workshop session
  Percentage of training course graduates who facilitated at least one workshop in the community within six months
Compliance with research assessed by completed surveys | through study completion, an average of 1 year
  Percentage of women who completed both baseline and post survey out of all participants
Proportion of participants who accept lay-led workshops, assessed by feedback forms | Last session of each workshop (workshops take place throughout one year)
  Workshop participants complete feedback forms self reporting on acceptability of duration and appropriateness of workshop content on a 1-5 Likert scale. Acceptability will include those who answered 4-5 on the Likert scale.
Proportion of participants satisfied with lay-led workshops, assessed by feedback forms | Last session of each workshop, (workshops take place throughout one year)
  Workshop participants complete feedback forms self reporting on overall satisfaction, satisfaction of workshop methods and satisfaction with facilitator on a 1-5 Likert scale. Satisfaction will include those who answered 4-5 on the Likert scale.

SECONDARY OUTCOMES:
Change in the level of food literacy | At baseline and three months after intervention
  Level of food literacy will be assessed by using a food literacy self report scale based on Poelman's Self-Perceived Food Literacy (SPFL) questionnaire, including 23 questions, score ranging between 23-65, the higher the score the higher the food literacy level.
Change in lay leaders' Self Efficacy: self report questionnaire | At baseline and three months after intervention
  Self Efficacy will be assessed through self report questionnaires (4 questions, 1-5 Likert scale), assessing participants self-efficacy in facilitating the food literacy material to target populations among trainers. The higher the average, the higher the self-efficacy.
Change in Mediterranean Diet adherence | At baseline and three months after intervention
  Women complete a validated self report survey, the Israel-Mediterranean Diet Adherence Screener (I-MEDAS) reporting on their adherence to the Mediterranean Diet, including consumption of sweets, sweet beverages, fruits and vegetables, whole grains, and legumes. The scale ranges between 1-17, the higher the score the higher the adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD, MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

REFERENCES:
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Desjardins, E.
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Kalter-Leibovici O, Chetrit A, Lubin F, Atamna A, Alpert G, Ziv A, Abu-Saad K, Murad H, Eilat-Adar S, Goldbourt U. Adult-onset diabetes among Arabs and Jews in Israel: a population-based study. Diabet Med. 2012 Jun;29(6):748-54. doi: 10.1111/j.1464-5491.2011.03516.x. PMID 22050554
- [Background] Vidgen HA, Gallegos D. Defining food literacy and its components. Appetite. 2014 May;76:50-9. doi: 10.1016/j.appet.2014.01.010. Epub 2014 Jan 22. PMID 24462490
- [Background] Wang H, Dwyer-Lindgren L, Lofgren KT, Rajaratnam JK, Marcus JR, Levin-Rector A, Levitz CE, Lopez AD, Murray CJ. Age-specific and sex-specific mortality in 187 countries, 1970-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2071-94. doi: 10.1016/S0140-6736(12)61719-X. PMID 23245603